CLINICAL TRIAL: NCT00151060
Title: Phase II Evaluation of Early Oral Estramustine, Oral Etoposide and Intravenous Paclitaxel in Patients With Hormonally Responsive Adenocarcinoma of the Prostate
Brief Title: Estramustine, Etoposide and Paclitaxel Treatment for Hormonally Responsive Adenocarcinoma of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9815
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estramustine; Etoposide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Estramustine, Etoposide and Paclitaxel (Experimental)
  Interventions: Drug: Estramustine; Drug: Etoposide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Estramustine
Drug: Etoposide
Drug: Paclitaxel

SUMMARY:
Hormonal therapy is the standard treatment for prostate cancer which has spread to other areas of the body. Despite the high initial response rates to hormonal therapy, the vast majority of men will develop cancer which is no longer responsive to hormone deprivation. The average time for hormonal therapy to be effective is about 18 months. Chemotherapy combinations which can treat the disease when it no longer responds to hormonal therapy have been developed, but these treatments are not curative. One of these combinations is estramustine, etoposide and paclitaxel. In men with far advanced disease, 60% will have a decrease in their PSA (Prostate Specific Antigen) or shrinkage of tumors after treatment with this chemotherapy. Despite this, these men have all developed further disease progression requiring additional treatment. One possible way to make chemotherapy more effective is to give it when the number of tumor cells is smallest, and the number of cells to be killed is at a low level. One situation in which this is true is when a man has responded to hormonal therapy any tumors are at their smallest size. This study will test whether the addition of chemotherapy at that time will prolong the time until the cancer becomes unresponsive to hormonal therapy.

ELIGIBILITY:
All patients must have a histologic diagnosis of adenocarcinoma of the prostate with evidence of metastases on bone or CT scan. Patients with regional metastases to pelvic lymph nodes (D1 disease) as their only site of metastases will be excluded from this study.

Patients on androgen suppression therapy at the time of registration must have received less than seven months of therapy (excluding any neoadjuvant hormonal therapy) and must have a decreasing or stable PSA level.

Patients may not be undergoing concurrent chemotherapy, biologic therapy, or radiation therapy. Prior to radiation therapy must have completed more than 4 weeks prior to registration.

Patients may not have received prior cytotoxic chemotherapy.

Patients may not have evidence of brain metastases or untreated spinal cord compression.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1998-12; Primary Completion 2004-11 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure | 4 Cycles
  Estimate the time to treatment failure in patients treated with combined androgen blockade and 4 cycles of estramustine, etoposide and paclitaxel.

CONTACTS AND LOCATIONS:
Overall Officials: David C. Smith, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer, Ann Arbor, Michigan, United States